CLINICAL TRIAL: NCT05642104
Title: The Detection of Cell-in-cell Structure (CICs) in Patients With Breast Cancer Undergoing Neoadjuvant Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Z211100002921033
Record Dates: First submitted 2022-11-02; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; cell-in-cell structures; Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Histopathological section
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group assignment: Patients with invasive breast cancer who need neoadjuvant therapy.
  Interventions: Drug: Neoadjuvant therapy

INTERVENTIONS:
Drug: Neoadjuvant therapy — all procedures is in accordance with international guidelines and domestic expert consensus on breast cancer.

SUMMARY:
Breast cancer is the most common malignant tumor in women worldwide and neoadjuvant therapy has been the standard care for local advanced breast cancer. Moreover, neoadjuvant therapy undoubtedly provides an ideal model to evaluate the response to therapy. Cell-in-cell structures (CICs) refer to the presence of one or more cells inside host cell, which generally leads to the death of inner cells. Notably, established evidences indicated that CICs were present in breast cancer and tend to impact patient survival. However, whether CICs profile could predict efficacy of therapy remains unclear. In this prospective cohort study, the CICs number and profile will be detected in tumor tissue before and after the neoadjuvant therapy. Then the association between CICs number including dynamic changing and response rate will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, female;
* Pathological biopsy confirmed invasive ductal carcinoma;
* Karnofsky Performance Status (KPS)≥ 60, expected survival ≥4 months;
* Locally advanced breast cancer (HER2-positive disease and TNBC, ≥cT1c or ≥cN0； HER2-negative，HR positive disease，≥cT2 or ≥cN1；Large primary tumor relative to breast size in a patient who desires breast conservation) ;
* According to the RECIST1.1 standard, at least one measurable lesion exists;

Exclusion Criteria:

* Pregnant or lactating women;
* Left ventricular ejection fraction less than 50%;
* History of malignant tumor and concurrent occurrence of other tumors;
* Serious medical pathology, such as congestive heart failure; unstable angina; uncontrolled high risk arrhythmias, and other serious illness or medical condition that may interfere with the study;
* Refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer treated with neoadjuvant therapy attending Beijing Shijitan Hospital from 2021-2023.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
pCR(complete pathological response) | Up to 24 weeks.
  no invasive malignant cells identifiable in sections from the site of the tumor（Miller-Payne grades 5） the Miller-Payne grades 4 and 5 patients are grouped as responders.
Objective response rate (ORR) | Up to 24 weeks.
  Response Evaluation Criteria in Solid Tumors (RECIST)：Progressive Disease (PD); Partial Response (PR); Complete Response (CR); Stable Disease (SD) Objective response rate (ORR), defined as the proportion of patients with a complete response (CR) partial response (PR) to treatment.
Quantification of CIC structure in tumor tissue | Up to 24 weeks.
  CICs number and subtypes in tumor tissue (Core needle biopsy specimens before and after neoadjuvant therapy and surgical specimens based on neoadjuvant therapy.)

OTHER OUTCOMES:
Disease-free survival (DFS) | Within 5 years after surgery
  It refers to the length of time from the start of medication after enrollment to the death of the patient because of the recurrence, distant metastasis of the disease, invasive contralateral breast cancer, or any other cause.
Overall survival (OS) | Within 10 years after surgery
  It refers to the length of time from the start of treatment to the death of the patient.
CEA(carcinoembryonic antigen) | Up to 24 weeks.
  Counts of international units per milliliter (IU/mL) of tumor marker CEA
CA125(Carbohydrate antigen125) | Up to 24 weeks.
  Counts of international units per milliliter (IU/mL) of tumor marker CA 125
CA199(Carbohydrate antigen199) | Up to 24 weeks.
  Counts of international units per milliliter (IU/mL) of tumor marker CA 199

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Huang, PHD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fais S, Overholtzer M. Cell-in-cell phenomena in cancer. Nat Rev Cancer. 2018 Dec;18(12):758-766. doi: 10.1038/s41568-018-0073-9. PMID 30420767
- [Background] Overholtzer M, Mailleux AA, Mouneimne G, Normand G, Schnitt SJ, King RW, Cibas ES, Brugge JS. A nonapoptotic cell death process, entosis, that occurs by cell-in-cell invasion. Cell. 2007 Nov 30;131(5):966-79. doi: 10.1016/j.cell.2007.10.040. PMID 18045538
- [Background] Galluzzi L, Vitale I, Abrams JM, Alnemri ES, Baehrecke EH, Blagosklonny MV, Dawson TM, Dawson VL, El-Deiry WS, Fulda S, Gottlieb E, Green DR, Hengartner MO, Kepp O, Knight RA, Kumar S, Lipton SA, Lu X, Madeo F, Malorni W, Mehlen P, Nunez G, Peter ME, Piacentini M, Rubinsztein DC, Shi Y, Simon HU, Vandenabeele P, White E, Yuan J, Zhivotovsky B, Melino G, Kroemer G. Molecular definitions of cell death subroutines: recommendations of the Nomenclature Committee on Cell Death 2012. Cell Death Differ. 2012 Jan;19(1):107-20. doi: 10.1038/cdd.2011.96. Epub 2011 Jul 15. PMID 21760595
- [Background] Schwegler M, Wirsing AM, Schenker HM, Ott L, Ries JM, Buttner-Herold M, Fietkau R, Putz F, Distel LV. Prognostic Value of Homotypic Cell Internalization by Nonprofessional Phagocytic Cancer Cells. Biomed Res Int. 2015;2015:359392. doi: 10.1155/2015/359392. Epub 2015 Oct 4. PMID 26504802
- [Background] Schenker H, Buttner-Herold M, Fietkau R, Distel LV. Cell-in-cell structures are more potent predictors of outcome than senescence or apoptosis in head and neck squamous cell carcinomas. Radiat Oncol. 2017 Jan 18;12(1):21. doi: 10.1186/s13014-016-0746-z. PMID 28100275
- [Background] Huang H, Chen A, Wang T, Wang M, Ning X, He M, Hu Y, Yuan L, Li S, Wang Q, Liu H, Chen Z, Ren J, Sun Q. Detecting cell-in-cell structures in human tumor samples by E-cadherin/CD68/CD45 triple staining. Oncotarget. 2015 Aug 21;6(24):20278-87. doi: 10.18632/oncotarget.4275. PMID 26109430
- [Background] Ruan B, Niu Z, Jiang X, Li Z, Tai Y, Huang H, Sun Q. High Frequency of Cell-in-Cell Formation in Heterogeneous Human Breast Cancer Tissue in a Patient With Poor Prognosis: A Case Report and Literature Review. Front Oncol. 2019 Dec 19;9:1444. doi: 10.3389/fonc.2019.01444. eCollection 2019. PMID 31921689
- [Background] Zhang X, Niu Z, Qin H, Fan J, Wang M, Zhang B, Zheng Y, Gao L, Chen Z, Tai Y, Yang M, Huang H, Sun Q. Subtype-Based Prognostic Analysis of Cell-in-Cell Structures in Early Breast Cancer. Front Oncol. 2019 Sep 20;9:895. doi: 10.3389/fonc.2019.00895. eCollection 2019. PMID 31681557